CLINICAL TRIAL: NCT05702840
Title: The Effects of a Home-based Resistance Training Programme on Body Composition and Muscle Function During Weight Loss in People With Overweight or Obesity: a Randomised Controlled Pilot Trial
Brief Title: EXerCise wEight Loss
Acronym: EXCEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Stuart Gray, Professor, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EXerCise wEight Loss Study
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Randomised controlled pilot trial with two groups, resistance exercise + weight loss group and weight loss only group.
Who Masked: Outcomes Assessor
Masking Description: Members of the research team that perform measurements are blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance exercise training + weight loss group (RT+WL) (Experimental): Participants (WL-RT) will be provided with a resistance exercise booklet containing instructions for exercises and links to demonstration videos. A demonstration and explanation of the exercises will be given at the beginning of the intervention, alongside a discussion of the principles of the programme such as starting level and progression. We will ask participants to perform the resistance exercises for 12-week period. Participants will be asked to perform exercises 3 times a week (3 sets reaching the RPE scale between 8 - 10 out of 10 (4-6 out of 10 in the first week)) for the intervention period. The exercises will include press-ups, band lateral raises, band seated low row, squat, lunge and calf raise.
  Interventions: Behavioral: Resistance exercise training + weight loss group
- Weight loss only group (WL) (Experimental): All participants (WL and WL-RT) will be provided with vouchers to access the weight watchers weight loss programme for a 12-week period. Weight Watchers is a commercially available programme and participants will set an initial goal to lose 5kg of body mass. If 5kg weight loss is achieved then the participant can chose further weight loss goals, as long as it would result in a body mass in the weight watchers healthy weight range (https://www.weightwatchers.com/uk/weight-loss/programme/tools/healthy-weight-chart).This plan works on the basis of an individualised points plan that can then be used by the participant to select foods/meals to consume throughout the day.
  Interventions: Behavioral: Weight loss only group (WL)

INTERVENTIONS:
Behavioral: Resistance exercise training + weight loss group — Doing resistance exercises as well as following the weight watchers weight loss programme for a 12-week period
  Arms: Resistance exercise training + weight loss group (RT+WL)
Behavioral: Weight loss only group (WL) — Only following the weight watchers weight loss programme for a 12-week period
  Arms: Weight loss only group (WL)

SUMMARY:
The overall aim of this study is to investigate the effects of home-based resistance exercise programme on changes in body composition and strength during weight loss, in people living with obesity or overweight.

ELIGIBILITY:
Inclusion Criteria:

* Obesity or overweight (BMI ≥ 25kg/m2).
* Passing the Physical Activity Readiness Questionnaire (PAR-q+)

Exclusion Criteria:

* Currently take part in more than 1.5 hours of structured exercise per week.
* Having recently (<6 months) taken part in any resistance exercise training, taking any medications known to affect weight loss.
* Actively engaged in a weight loss programme, having lost more than 2kg weight in the last 6 months.
* Any other reason which would limit ability to perform the exercises and outcome measurements safely.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in whole body lean mass | Change from baseline to 12 weeks
  whole body lean mass measured via bio-electrical impedance

SECONDARY OUTCOMES:
Change in whole body fat mass | Change from baseline to 12 weeks
  whole body fat mass measured via bio-electrical impedance
Change in body mass | Change from baseline to 12 weeks
  body mass measured on scales
Change in vastus lateralis muscle thickness | Change from baseline to 12 weeks
  Muscle thickness of the vastus lateralis muscle measured via ultrasound
Change in knee extensor maximal isometric torque | Change from baseline to 12 weeks
  Knee extensor maximal isometric torque measured during a maximal voluntary contraction
Change in grip strength | Change from baseline to 12 weeks
  Grip strength measured with a hand held dynamometer
Change in functional physical abilities | Change from baseline to 12 weeks
  A 30-second sit-to-stand test measured functional abilities

CONTACTS AND LOCATIONS:
Locations (1):
- Stuart Robert Gray, Glasgow, United Kingdom

REFERENCES:
- [Background] Upadhyay J, Farr O, Perakakis N, Ghaly W, Mantzoros C. Obesity as a Disease. Med Clin North Am. 2018 Jan;102(1):13-33. doi: 10.1016/j.mcna.2017.08.004. Epub 2017 Oct 21. PMID 29156181
- [Background] An R, Ji M, Zhang S. Global warming and obesity: a systematic review. Obes Rev. 2018 Feb;19(2):150-163. doi: 10.1111/obr.12624. Epub 2017 Oct 4. PMID 28977817
- [Background] James PT, Leach R, Kalamara E, Shayeghi M. The worldwide obesity epidemic. Obes Res. 2001 Nov;9 Suppl 4:228S-233S. doi: 10.1038/oby.2001.123. PMID 11707546
- [Background] Siervo M, Montagnese C, Mathers JC, Soroka KR, Stephan BC, Wells JC. Sugar consumption and global prevalence of obesity and hypertension: an ecological analysis. Public Health Nutr. 2014 Mar;17(3):587-96. doi: 10.1017/S1368980013000141. Epub 2013 Feb 18. PMID 23414749
- [Background] Ge L, Sadeghirad B, Ball GDC, da Costa BR, Hitchcock CL, Svendrovski A, Kiflen R, Quadri K, Kwon HY, Karamouzian M, Adams-Webber T, Ahmed W, Damanhoury S, Zeraatkar D, Nikolakopoulou A, Tsuyuki RT, Tian J, Yang K, Guyatt GH, Johnston BC. Comparison of dietary macronutrient patterns of 14 popular named dietary programmes for weight and cardiovascular risk factor reduction in adults: systematic review and network meta-analysis of randomised trials. BMJ. 2020 Apr 1;369:m696. doi: 10.1136/bmj.m696. PMID 32238384
- [Background] Lean ME, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Stefanetti R, Trenell M, Welsh P, Kean S, Ford I, McConnachie A, Sattar N, Taylor R. Primary care-led weight management for remission of type 2 diabetes (DiRECT): an open-label, cluster-randomised trial. Lancet. 2018 Feb 10;391(10120):541-551. doi: 10.1016/S0140-6736(17)33102-1. Epub 2017 Dec 5. PMID 29221645
- [Background] Cava E, Yeat NC, Mittendorfer B. Preserving Healthy Muscle during Weight Loss. Adv Nutr. 2017 May 15;8(3):511-519. doi: 10.3945/an.116.014506. Print 2017 May. PMID 28507015
- [Background] Enriquez Guerrero A, San Mauro Martin I, Garicano Vilar E, Camina Martin MA. Effectiveness of an intermittent fasting diet versus continuous energy restriction on anthropometric measurements, body composition and lipid profile in overweight and obese adults: a meta-analysis. Eur J Clin Nutr. 2021 Jul;75(7):1024-1039. doi: 10.1038/s41430-020-00821-1. Epub 2020 Dec 9. PMID 33293678
- [Background] Pellegrini M, Cioffi I, Evangelista A, Ponzo V, Goitre I, Ciccone G, Ghigo E, Bo S. Effects of time-restricted feeding on body weight and metabolism. A systematic review and meta-analysis. Rev Endocr Metab Disord. 2020 Mar;21(1):17-33. doi: 10.1007/s11154-019-09524-w. PMID 31808043
- [Background] Wolfe RR. The underappreciated role of muscle in health and disease. Am J Clin Nutr. 2006 Sep;84(3):475-82. doi: 10.1093/ajcn/84.3.475. PMID 16960159
- [Background] Sajoux I, Lorenzo PM, Gomez-Arbelaez D, Zulet MA, Abete I, Castro AI, Baltar J, Portillo MP, Tinahones FJ, Martinez JA, Crujeiras AB, Casanueva FF. Effect of a Very-Low-Calorie Ketogenic Diet on Circulating Myokine Levels Compared with the Effect of Bariatric Surgery or a Low-Calorie Diet in Patients with Obesity. Nutrients. 2019 Oct 4;11(10):2368. doi: 10.3390/nu11102368. PMID 31590286
- [Background] Ashton RE, Tew GA, Aning JJ, Gilbert SE, Lewis L, Saxton JM. Effects of short-term, medium-term and long-term resistance exercise training on cardiometabolic health outcomes in adults: systematic review with meta-analysis. Br J Sports Med. 2020 Mar;54(6):341-348. doi: 10.1136/bjsports-2017-098970. Epub 2018 Jun 22. PMID 29934430
- [Background] Cornelissen VA, Fagard RH, Coeckelberghs E, Vanhees L. Impact of resistance training on blood pressure and other cardiovascular risk factors: a meta-analysis of randomized, controlled trials. Hypertension. 2011 Nov;58(5):950-8. doi: 10.1161/HYPERTENSIONAHA.111.177071. Epub 2011 Sep 6. PMID 21896934
- [Background] Plotnikoff RC, Eves N, Jung M, Sigal RJ, Padwal R, Karunamuni N. Multicomponent, home-based resistance training for obese adults with type 2 diabetes: a randomized controlled trial. Int J Obes (Lond). 2010 Dec;34(12):1733-41. doi: 10.1038/ijo.2010.109. Epub 2010 Jun 8. PMID 20531348
- [Background] Mikesky AE, Topp R, Wigglesworth JK, Harsha DM, Edwards JE. Efficacy of a home-based training program for older adults using elastic tubing. Eur J Appl Physiol Occup Physiol. 1994;69(4):316-20. doi: 10.1007/BF00392037. PMID 7851367
- [Background] Zion AS, De Meersman R, Diamond BE, Bloomfield DM. A home-based resistance-training program using elastic bands for elderly patients with orthostatic hypotension. Clin Auton Res. 2003 Aug;13(4):286-92. doi: 10.1007/s10286-003-0117-3. PMID 12955554
- [Background] NIH Consensus statement. Bioelectrical impedance analysis in body composition measurement. National Institutes of Health Technology Assessment Conference Statement. December 12-14, 1994. Nutrition. 1996 Nov-Dec;12(11-12):749-62. PMID 8974099
- [Derived] Binmahfoz A, Johnston L, Dunning E, Gray CM, Gray SR. The effects of a home-based resistance training programme on body composition and muscle function during weight loss in people living with overweight or obesity: a randomised controlled pilot trial. Nutr Metab (Lond). 2025 Aug 4;22(1):90. doi: 10.1186/s12986-025-00986-1. PMID 40760444